CLINICAL TRIAL: NCT01958294
Title: The MICHI NEUROPROTECTION SYSTEM: Evaluation of Performance in Carotid Artery Stent Procedures (The LOTUS Study)
Acronym: LOTUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Silk Road Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRM-2011-01
Record Dates: First submitted 2013-10-04; First posted 2013-10-09 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-03

CONDITIONS: Carotid Stenosis; Carotid Artery Disease
MeSH Terms: conditions — Carotid Stenosis; Carotid Artery Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MICHI Neuroprotection System (Other): Subjects enrolled into this study will be male or female subjects who are candidates for carotid angioplasty and stenting, who, after meeting all of the eligibility criteria, undergo transcervical Carotid Artery Stenting with carotid flow reversal using the MICHI Neuroprotection System.
  Interventions: Device: MICHI Neuroprotection System

INTERVENTIONS:
Device: MICHI Neuroprotection System
  Other Names: MICHI NPS; MICHI NPS + f

SUMMARY:
The LOTUS Study is intended to demonstrate the usability of the MICHI Neuroprotection System (MICHI NPS) or MICHI Neuroprotection System with filter (MICHI NPS+f) for use in subjects who are candidates for Carotid Artery Stenting (CAS). It is a prospective, single arm study in which a maximum of 30 study subjects, and a run-in enrollment of up to 10 subjects will be followed immediately post-op and at 30 days.

DETAILED DESCRIPTION:
Cerebral embolization during carotid artery stenting (CAS) can often precipitate severe adverse neurological effects. Most major clinical studies of CAS have used distal filters for cerebral protection and have compared the neurologic complication rates with those of carotid endarterectomy (CEA). Many currently available embolic protection devices, however, have limited efficacy in capturing microembolic debris liberated during stenting, pre-dilatation and post-dilatation. Furthermore, distal protection systems are limited by the need to cross the lesion prior to deployment. Some studies have shown a relatively high incidence of cerebral infarction even when distal protection devices are employed.

Cerebral protection with carotid flow reversal is a method that was developed by Parodi, et al. (2005), as an alternative to the use of distal protection devices. While novel in its approach, this method too has its limitations. Criado, et al. (2004), developed a derivative technique that employs carotid flow reversal prior to traversing the stenosis that can be accomplished by directly accessing carotid anatomy without the use of the transfemoral approach. Major benefits to this method include the ability to perform the procedure on patients with severe carotid tortuosity and difficult aortic arch anatomy.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be > 21 years of age.
* Subject has the ability to understand and cooperate with study procedures and agrees to return for all required follow-up visits, tests, and exams.
* International Normalized Ratio (INR) must be ≤ 1.5 at the time of the procedure (subjects taking warfarin may be included if their dose is tapered prior to the procedure to meet the inclusion criterion. Dose may be returned to a therapeutic level after the procedure).
* The subject must sign a written informed consent prior to the procedure, using a form that is approved by the local medical Ethics Committee (EC).
* The life expectancy of the subject is at least one year.
* The subject has a lesion located in the internal carotid artery (ICA); the carotid bifurcation may be involved.
* The subject must have a minimum distance of 5 cm between the clavicle and bifurcation, as assessed by duplex Doppler ultrasound, computed axial tomographic (CT) angiography or magnetic resonance (MR) angiography.

Exclusion Criteria:

* The subject is participating in another investigational study that would interfere with the conduct or result of this study.
* The subject has dementia or a neurological illness that may confound the neurological evaluation.
* Presence of any one of the following anatomic risk factors:

  * Previous radiation treatment to the neck or radical neck dissection
  * Tracheostomy or tracheal stoma
  * Laryngectomy
  * Contralateral laryngeal nerve palsy
  * Severe tandem lesions
  * Inability to extend the head due to cervical arthritis or other cervical disorders
* Total occlusion of the target vessel.
* There is an existing, previously placed stent in the target artery.
* The subject has a known life-threatening allergy to the contrast media that cannot be treated.
* Subject has history of intolerance or allergic reaction to any of the study medications including aspirin, clopidogrel bisulfate (Plavix®) or ticlopidine (Ticlid®), prasugrel heparin or bivalirudin (Angiomax™). Subjects must be able to tolerate a combination of aspirin and clopidogrel/ticlopidine or prasugrel.
* The subject has a gastrointestinal bleed that would interfere with antiplatelet therapy.
* The subject has known cardiac sources of emboli.
* Subject has Hemoglobin (Hgb) less than 8 gm/dL (unless on dialysis), platelet count < 50,000/mm3, or known heparin associated thrombocytopenia.
* Subject has documented atrial fibrillation in the prior 90 days.
* The subject has a history of bleeding diathesis or coagulopathy including thrombocytopenia or an inability to receive heparin in amounts sufficient to maintain an activated clotting time (ACT) at > 250, or if the subject will refuse blood transfusions.
* The subject has atherosclerotic disease involving the ipsilateral common carotid artery (CCA) that precludes safe placement of the sheath.
* The subject has abnormal angiographic findings other than that of the target lesion that indicate the subject is at risk for a stroke, such as: ipsilateral arterial stenosis greater in severity than the target lesion, cerebral aneurysm, or arteriovenous malformation of the cerebral vasculature.
* There is evidence of a carotid artery dissection prior to the initiation of the procedure.
* There is an angiographically visible thrombus.
* There is any condition that precludes proper angiographic assessment or makes percutaneous arterial access unsafe, e.g. morbid obesity, sustained systolic blood pressure > 180 mm Hg, tortuosity, occlusive disease, vessel anatomy or aortic arch anatomy.
* Occlusion (TIMI 0 flow), or string sign of the ipsilateral common or internal carotid artery.
* There is evidence of bilateral carotid stenosis that would require intervention within 30 days of procedure.
* There is evidence of a major stroke (NIHSS ≥10) within the previous 30 days of the procedure or the patient is considered, by the investigator, to be at high risk for hemorrhagic stroke.
* There is a planned treatment of a non-target lesion within 30 days post procedure.
* There is a history of intracranial hemorrhage within the previous 3 months, including hemorrhagic transformation of an ischemic stroke.
* There is history of an ipsilateral stroke with fluctuating neurologic symptoms within one year prior to the procedure.
* Female subjects who are pregnant (negative pregnancy test is required in women of childbearing potential).
* Subjects, who the Investigator determines, to be at risk of Deep Vein Thrombosis (DVT)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-08; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sumaira Macdonald, FRCP FRCR PhD EBIR, Principal Investigator — Newcastle upon Tyne Hospitals NHS Foundation Trust
Locations (1):
- Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, England, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- MICHI Neuroprotection System: Subjects enrolled into this study will be male or female subjects who are candidates for carotid angioplasty and stenting, who, after meeting all of the eligibility criteria, undergo transcervical Carotid Artery Stenting with carotid flow reversal using the MICHI Neuroprotection System.
  MICHI Neuroprotection System The MICHI Neuroprotection System (MICHI NPS) is a flow reversal circuit consisting of two proprietary sheaths connected by standard surgical tubing. The sheaths each have a standard hemostasis valve and sidearm. An in-line flow regulator allows the clinician to modify the flow through the circuit (either high flow or low flow) in addition to permitting temporary cessation of flow.
  The system permits transcervical access to the carotid lesion, and the flow reversal through the circuit re-directs emboli that are liberated during carotid angioplasty and stent delivery.
Period: Overall Study
Arm/Group | MICHI Neuroprotection System
Started | 12
Completed | 10
Not Completed | 2
Not completed — Clinical Circumstances | 2

BASELINE CHARACTERISTICS:
Population: Enrolled patients with extracranial carotid stenosis who were candidates for angioplasty and Carotid Artery Stenting.
Groups:
- MICHI Neuroprotection System: Subjects enrolled into this study will be male or female subjects who are candidates for carotid angioplasty and stenting, who, after meeting all of the eligibility criteria, undergo transcervical Carotid Artery Stenting with carotid flow reversal using the MICHI Neuroprotection System.
  MICHI Neuroprotection System
Arm/Group | MICHI Neuroprotection System
Number analyzed (Participants) | 12
Age, Customized [Number; unit: participants]
  70-74 years of age | 8
  75-79 years of age | 2
  80 years of age and older | 1
  Unknown or not reported | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 12
Average Height [Mean (Standard Deviation); unit: cm] | 163.8 (7.4)
Average Weight [Mean (Standard Deviation); unit: kg] | 71.7 (12.7)

OUTCOME MEASURES:

1. Primary Outcome: Composite of Any Stroke, Myocardial Infarction and Death
Description: Composite Major Adverse Event (MAE) Rate of any stroke, myocardial infarction and death during the 30-day post procedural period.
Time Frame: 30-days post-procedurally
Population: Composite Major Adverse Event (MAE) Rate of any stroke, myocardial infarction and death during the 30-day post procedural period.
Measure: Number; unit: participants
Arm/Group | MICHI Neuroprotection System
Number analyzed (Participants) | 10
participants
  Myocardial Infarction | 1
  Stroke | 0
  Death | 0

2. Secondary Outcome: Acute Device Success
Description: Acute device success - Defined as MICHI™ NPS was delivered (vascular access achieved), reverse flow was attempted and established and the device retrieved / removed from vasculature.
Time Frame: Intra procedural (1 day)
Population: Subjects meeting the description of the outcome measures in which vascular access was achieved, reverse flow was successfully established, and the device retrieved from the vasculature.
Measure: Number; unit: participants
Arm/Group | MICHI Neuroprotection System
Number analyzed (Participants) | 10
participants | 10

3. Secondary Outcome: Procedural Success
Description: Procedure Success - Procedural success is the ability to deliver therapeutic devices (balloons, stents, etc.) through the Transcervical Arterial Sheath and the ability to provide embolic protection throughout the procedure with the freedom of device related Major Adverse Events at 30 days.
Time Frame: Through 30-day Follow-up period
Population: Successful delivery of therapeutic devices (balloons, stents, etc.) through the Transcervical Arterial Sheath and ability to provide embolic protection throughout the procedure with freedom from device related Major Adverse Events at 30 days
Measure: Number; unit: participants
Arm/Group | MICHI Neuroprotection System
Number analyzed (Participants) | 10
participants | 9

ADVERSE EVENTS:
Time Frame: 0 to 30 days following study index procedure
Description: The protocol's primary endpoint was to capture MAEs, or Major Adverse Events, which differ from the ClinicalTrials.gov definition of Serious Adverse Events in that they only include Myocardial Infarction, Stroke and Death as determined by a Central Adjudication Committee (CEC), however, despite this difference, MAEs, SAES and AEs were all captured for documentation and data purposes.
Arm/Group | MICHI Neuroprotection System
Serious Adverse Events (participants affected / at risk) | 2/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MICHI Neuroprotection System (N=12)
Hematoma (Vascular disorders) | 2 (2) — SAEs were not reviewed by the independent Clinical Events Committee (CEC) because no MI Stroke or Death. Neither of these events was deemed to be related to the study device.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MICHI Neuroprotection System (N=12)
Bradycardia (Cardiac disorders) | 1 (1)
Dyspnea (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Indigestion (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Swelling (General disorders) | 1 (1)
Procedural Complication (Transient Intolerance) (Injury, poisoning and procedural complications) | 1 (1)
Vascular Procedure Complication (Injury, poisoning and procedural complications) | 1 (1)
Blood Troponin, CK or CK-MB Increased (Investigations) | 2 (2)
Full Blood Count Abnormal (Investigations) | 2 (2)
Hemoglobin Decreased (Investigations) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Right Arm Drift (Nervous system disorders) | 1 (1)
Transient Ischemic Attack (Nervous system disorders) | 1 (1)
Hematoma (Vascular disorders) | 6 (6)
Hemorrhage/Oozing (Vascular disorders) | 6 (6)
Hypertension (Vascular disorders) | 4 (4)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less